CLINICAL TRIAL: NCT00173108
Title: Early Intervention for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other); National Health Research Institutes, Taiwan (Other)
Responsible Party: Suh-Fang, Jeng, School and Graduate Insistute of Physical Therapt, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 9461700406
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: Premature Birth
Keywords: Prematurity; Early intervention; Neurodevelopment; Cost-effectiveness
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Term group (No Intervention)
- Usual care program group (No Intervention)
- Clinic-based interveniton program group (Experimental)
  Interventions: Behavioral: clinic-based intervention program and home-based intervention program
- Home-based interveniton program group (Experimental)
  Interventions: Behavioral: clinic-based intervention program and home-based intervention program

INTERVENTIONS:
Behavioral: clinic-based intervention program and home-based intervention program — The intervention includes education of child development skills, health and feeding consultation, intervention of mother-infant interaction, and parent support. Clinic-based intervention program is delivered in clinic while home-based intervention program is delivered at home.
  Arms: Clinic-based interveniton program group; Home-based interveniton program group

SUMMARY:
The first aim is to develop a clinic-based intervention program and a home-based intervention program for VLBW preterm infants that have common intervention services but are respectively delivered at clinic and home. The interventions are comprehensive that combine child- and parent-focused services including health and feeding consultation, education of child development skills, intervention of mother-infant interaction, and parent support. The eleven-session interventions are intensive that begin in hospitalization and end at 12 months of corrected age. The clinical feasibility and usefulness of implementing these intervention programs within the context of randomized intervention study subject to the existing constraints of the hospital and home settings will be tested in a pilot study.

The second aim is to conduct a randomized control trial to examine the costs and effectiveness of the UCP, the CBIP, and the HBIP for VLBW preterm infants. Gender and socio-economically matched normal full-term infants will also be included as a comparison group. Outcome measures that include child, parenting, and transactions outcomes will be compared between groups. Child outcome measures will include health status, growth, neurodevelopment, and neurosensory status; parenting outcome measures will include maternal parenting competence, social support, and psychological stress; transactions outcome measure will be mother-infant interaction. Costs (direct and indirect costs) associated with each early intervention program during the follow-up period will be estimated. Average and incremental cost/effectiveness ratio will be calculated to determine which early intervention program is most cost-effective for VLBW preterm infants.

DETAILED DESCRIPTION:
Preterm birth with very low birth weight (VLBW) (gestational age <37 weeks and birth weight <1,501 g) is a significant public health problem worldwide. Longitudinal follow-up studies showed that VLBW preterm infants require prolonged hospitalization and are at substantial risk for various morbidities during neonatal period than those born at normal birth weight. Furthermore, approximately 40% of VLBW preterm infants are burden with adverse outcomes from chronic health problems and re-hospitalizations, to lower IQ, developmental delays, behavioral problems, and poor educational achievement. Accumulating data collected in Western developed countries have suggested that comprehensive and intensive early interventions may be beneficial for preterm infants and their families. However, there is little information concerning what early intervention should be attempted for these infants and their families in Taiwan. The purpose of this study is therefore to examine the cost-effectiveness of three early intervention programs i.e., the usual care program, the clinic-based intervention program, and the home-based intervention program for VLBW preterm infants. In a preliminary study, we surveyed the need of intervention services following hospital discharge in VLBW preterm infants (N=69) and their families. All mothers expressed the need of services that 60 (87%) preferred service delivery at home and 9 (13%) preferred service delivery at neonatal follow-up clinic. The intervention services specifically identified were health and respiratory assistance (N=22), feeding assistance (N=17), education of child development skills (N=12), and parent support (N=8). Based on these survey data and the results of previous intervention studies, we will develop in this proposed research project a clinic-based intervention program and a home-based intervention program that have common intervention services but are respectively delivered via clinic visit and home visit. The interventions are comprehensive that combine child- and parent-focused services including health and feeding consultation, education of child development skills, intervention of mother-infant interaction, and parent support. The eleven-session interventions are intensive that begin in hospitalization and end at 12 months of corrected age.

This will be a four-year research project that employs a single blind, randomized experimental design to examine the efficacy of the early intervention programs for VLBW preterm infants. For the first year, we will develop the clinic-based intervention program and the home-based intervention programs in the actual situations to examine their clinical usefulness. From the second to the fourth year, 180 VLBW preterm infants who are born and admitted to the neonatal intensive care units of National Taiwan University Hospital and MacKay Memorial Hospital will be randomly assigned to the usual care program, the clinic-based intervention program, and the home-based intervention program. Sixty gender and socio-economically matched normal full-term infants will also be included as a comparison group. Child, parenting, and transactions outcomes will be assessed when infants are at 4, 6, 12, 18, and 24 months of corrected age. Child outcomes are measured by health status, growth, neurodevelopment, and neurosensory status; parenting outcomes are measured by maternal parenting competence, social support, and psychological stress; transactions outcome is measured by mother-infant interaction. Generalized estimating equations will be used to examine the differences in changes of outcome variables between intervention and control groups. At the end of the fourth year, the costs and effectiveness of the three intervention programs will be compared to determine which one is more cost-effective for VLBW preterm infants in Taiwan. The results of this study will help clinicians and parents understand the efficacy of early intervention for VLBW preterm infants. Furthermore, the data of this study will provide important information to policy makers and health administrators concerning resource allocation of early intervention forVLBW preterm infants in Taiwan.

ELIGIBILITY:
Inclusion Criteria for preterm infants:

* BW below 1,501 gm
* GA under 37 weeks
* Admission to the NICU within the first 7 days of life
* Physiologically stable at PCA 36 weeks as diagnosed by attending physician
* Hospital discharge prior to PCA 40 weeks
* Absence of congenital anomalies and/or severe neonatal diseases
* Family residence in the greater Taipei area.

Exclusion Criteria for preterm infants:

* Severe neonatal diseases included major neurologic abnormalities (such as seizures, hydrocephalus, ventriculoperitoneal shunt, meningitis, periventricular leukomalacia, grade III-IV intraventricular hemorrhage, and grade IV retinopathy of prematurity)
* Necrotizing enterocolitis with colostomy
* Severe cardiopulmonary disease requiring daily oxygen use at hospital discharge

Inclusion Criteria for full-term infants:

* Birth weight >2,500 g;
* Gestational age within 38-42 weeks,
* Family living in the same geographic region as those of the VLBW preterm infants

Exclusion Criteria for full-term infants:

* Serious prenatal or perinatal complications

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2006-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Compare the costs and effectiveness of the three intervention programs to determine which one is more cost-effective for VLBW preterm infants in Taiwan. | In-hospital, 6, 12, 18 and 24 months of age
  Effectiveness includes the child (health, growth, neurodevelopment, and neurosensory), parent (competence, social support, and psychological stress) and transaction outcomes (parent-child interaction). Cost includes direct and indirect cost related to health and intervention program

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Sc.D, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Derived] Li SJ, Tsao PN, Tu YK, Hsieh WS, Yao NJ, Wu YT, Jeng SF. Cognitive and motor development in preterm children from 6 to 36 months of age: Trajectories, risk factors and predictability. Early Hum Dev. 2022 Sep;172:105634. doi: 10.1016/j.earlhumdev.2022.105634. Epub 2022 Jul 28. PMID 35921693
- [Derived] Su YH, Jeng SF, Hsieh WS, Tu YK, Wu YT, Chen LC. Gross Motor Trajectories During the First Year of Life for Preterm Infants With Very Low Birth Weight. Phys Ther. 2017 Mar 1;97(3):365-373. doi: 10.1093/ptj/pzx007. PMID 28339607
- [Derived] Wu YC, Leng CH, Hsieh WS, Hsu CH, Chen WJ, Gau SS, Chiu NC, Yang MC, Li-Jung Fang, Hsu HC, Yu YT, Wu YT, Chen LC, Jeng SF. A randomized controlled trial of clinic-based and home-based interventions in comparison with usual care for preterm infants: effects and mediators. Res Dev Disabil. 2014 Oct;35(10):2384-93. doi: 10.1016/j.ridd.2014.06.009. Epub 2014 Jun 26. PMID 24973546